Study ID:IRB202001790 Date Approved: 11/1/2023

NCT04705363





## Institutional Review Board Health Science Center

**Title of Project**: A sociolinguistic-enabled web application to develop precision health intervention for African

Americans

Principal Investigator: Melissa Vilaro PhD, Assistant Professor in Health and Wellness

Department of Family, Youth and Community Sciences

University of Florida | IFAS

- 1. **Purpose of the Study:** This study is being done to help build virtual health assistants (VHA) that work better for patients who are between the ages of 45 and 75 and may be in need of a colorectal cancer (CRC) screening. A VHA is a digital healthcare professional designed to help patients like you better understand the importance and procedures of CRC screenings. Past studies have shown that VHAs make the patient feel much more at ease and confident in the healthcare advice and assistance offered. In this study, you will interact with a VHA who will explain the importance and procedures of CRC screenings. You will then be asked your opinion of the interaction and of the VHA. Your responses will help the researchers better understand how to improve the VHAs in order to benefit patients to the fullest.
- 2. **Procedures to be followed:** You will be randomly assigned (much like the flip of a coin) by a computer program to interact with one of two possible VHAs. One VHA will be a computer-generated doctor who will have a conversation with you. The other possible VHA will consist of photos of the computer-generated doctor with text that will guide you through the interaction. If you take part in this study, you will be offered a detailed explanation of CRC screenings and the benefits they offer you through interaction with the VHA. You will then be asked to take a survey to give your opinion of your experience with the VHA.
- 3. **Duration:** Your interaction with the VHA through the survey should take less than an hour.
- 4. **Research Benefits:** There are no direct benefits from participating in this study. However, you may gain important information on your individual risk of developing colorectal cancer. You will also learn how to screen for colorectal cancer.
- 5. **Research Risks:** There may be some possibility of mild emotional discomfort from being presented potential risks of a disease. However, the probability of any physical, mental, or social harm is little to none.
- 6. **Statement of Confidentiality:** Your participation in this research is confidential. The survey does not ask for any information that would identify who the responses belong to. In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared because your name is in no way linked to your responses. The data collected from your participation in this study will be held in Dropbox, a file sharing system approved by UF Integrated Risk Management. The data collected will include your responses to survey questions and information about your interactions with the intervention.

Study ID:IRB202001790 Date Approved: 11/1/2023



- 7. **Right to Ask Questions:** You may contact Dr. Melissa Vilaro at 352-273-3525 at any time if you have questions about the research or if you think that you have been hurt by the research. You may contact the Institutional Review Board at the University of Florida Health Science Center at (352) 273-9600 if you have questions about your rights as a research subject or what to do if you are injured.
- 8. **Payment for participation:** You will receive \$6 compensation for your participation. The panel company you are working with will arrange payment once you have finished the survey.
- 9. **Cost:** There is no cost to participating in this study.
- 10. **Voluntary Participation:** Your decision to be in this research is voluntary. You may choose not to participate in this study. If you choose to participate, you may quit the study at any time after you have begun and there will be no penalty and no loss of any benefits you are entitled to. If any new findings related to the communication and/or guidelines of CRC screening become available and affect your participation, you will be told.
- 11. **Clinicaltrials.gov:** A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Completion and return of the survey implies that you have read the information in this form and consent to take part in the research. Please keep this form for your records or future reference.